CLINICAL TRIAL: NCT03431285
Title: Ketamine for Acute Painful Crisis in Sickle Cell Disease Patients: Prospective Randomized Control Trial
Brief Title: Ketamine for Acute Painful Crisis in Sickle Cell Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Mohammed Saeed Saad Alshahrani, Associate professor - Emergency medicine, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR3- 2017-01- 192
Record Dates: First submitted 2018-02-07; First posted 2018-02-13 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Crisis
MeSH Terms: conditions — Vaso-Occlusive Crises | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple-blind study. The study solution will be prepared in identical 100-ml Normal Saline bags by the research nurse
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphine Group (Active Comparator): Patients will receive standard dose of morphine (0.1 mg/kg) in 100 ml normal saline (NS) infused over 30 minutes in addition to standard IV hydration.
  Interventions: Drug: Morphine Group; Other: standard IV hydration
- Ketamine Group (Active Comparator): Patients will receive low dose ketamine 0.3 mg/kg in 100ml normal saline (NS) infused over 30 minutes in addition to standard IV hydration
  Interventions: Drug: Ketamine Group; Other: standard IV hydration

INTERVENTIONS:
Drug: Morphine Group — Patients will receive standard dose of morphine (0.1 mg/kg) in 100 ml normal saline infused over 30 min in addition to standard IV hydration.
  Other Names: Control Group
  Arms: Morphine Group
Drug: Ketamine Group — Patients will receive low dose ketamine 0.3 mg/kg in 100ml N.S. infused over 30 min in addition to standard IV hydration
  Other Names: Intervention Group
  Arms: Ketamine Group
Other: standard IV hydration — IV hydration as per our institutional protocol (Lactated Ringer's or NaCl 0.9% solution will be infused at a rate of 2-3 ml/kg/h)

SUMMARY:
Investigators hypothesize that administration of ketamine for pain relief in sickle cell patients with vaso-occlusive crisis early on will lead to a more rapid improvement in pain score and less narcotic requirement.

DETAILED DESCRIPTION:
Sickle cell disease is an inherited hematological disorder where the shape of red blood cells (RBC) is altered into a sickle-like cells resulting in red blood cell destruction and therefore anemia and other complications. It's a widely spread condition in African American population as well as the Southern and Eastern Provinces of Arabian Peninsula.

Acute painful episodes are a very common complication of the disease process, mainly thought to be a result of tissue ischemia due to occlusion of the microcirculation with clusters of sickled RBC(1). This usually involves long bones or spine but can involve other areas. Acute painful crises can also be precipitated by cold exposure, dehydration, infection, hypoxia, acidosis, hypercarbia, or in some cases it is not related to a specific trigger. This condition puts the patient in severe pain requiring multiple Emergency Department (ED) visits and sometimes admission to the hospital. Currently the mainstay of therapy for acute painful crises is hydration and IV analgesia (2). This makes pain control challenging for the emergency physician as management of acute painful crises requires multiple doses of intravenous (IV) opioids. A retrospective study of 19 patients and 57 visits showed that accumulative dose of IV morphine ranged between 4 milligram (mg) and 26.7 (0.05-0.5 mg/kg) during 70% of the visits. 50% of the patients were admitted after less than 3 hours of ED treatment, 28% of the discharged patients returned to the ED within 3 days (3). Also, as other chronic pain patients, sickle cell disease patients develop opioid induced hyperalgesia (OIH) leading to activation of N- methyl D Aspartate receptors (NMDA) (1).

The use of ketamine, a non-competitive NMDA receptor antagonist, may have the potential to modulate the OIH through impaired sensitization of spinal neurons to nociceptive stimuli and may, therefore, impede development of and blunt neuropathic pain. Extensive search of literature databases showed few published reports and retrospective studies including few patients which have addressed the use of low-dose ketamine in the management of acute painful crises in sickle cell disease (SCD) (4-6). A retrospective study (5) included 5 children and adolescents received a low-dose ketamine infusion for the treatment of sickle cell-related pain demonstrated reduced pain scores in 40% of patients and significant reduction in opioid utilization in only 20% of patients. However, that report was retrospective in nature, non-powered, and included few patients. A recent Canadian retrospective study including 9 adult and adolescent patients demonstrated statistically significant reduced cumulative morphine consumption (146±16.5 mg/day vs. 112.±12.2 mg/day) and pain scores after adding intravenous ketamine in patients with painful sickle cell crises (7). Similarly, another American investigators reported decreased opioid consumption with infusing low-dose ketamine as an adjuvant analgesic in 30 patients presented with sickle cell disease with vaso-occlusive crisis (VOC), that study was retrospective (2). Moreover, in year 2017, a prospective, randomized, double dummy trial was done comparing the adverse effects and analgesic efficacy of low-dose ketamine for acute pain in the ED either by single intravenous push or short infusion. This study shows that low-dose ketamine administered as short infusion is related with a significantly lower rates of feeling of unreality and sedation with no difference in analgesic efficacy in comparison to intravenous push (8)

To the best of investigator's knowledge, there is no large, prospective, comparative, controlled clinical trial investigated in the addition of low-dose ketamine in shortening the ER stays and improving the quality of analgesia in patients with VOC.

Sample Size

A data obtained from a pilot study included 10 patients who received either morphine or ketamine showed that the mean and SD of pain visual analogue score (VAS) at 1-hour following administering the study drug among patients presented with sickle-cell VOC were (Morphine 6.5 ± 3.41565, Ketamine: 1.6667 ± 1.52753).

An a priori power analysis indicated that a sample size of 220 patients is sufficiently large to detect a mean difference in the pain VAS of 1.5 that would have a clinical importance, with a type-I error of 0.05 and a power of 90%. Additional patients (20%) will be added for a final sample size of 264 patients to compensate for those dropping out during the study.

Interim Analysis

An independent safety committee will perform three interim analyses on information time 25% (55 patients), 50% (110 patients) and 75% (165 patients). Data evaluation at each interim analysis will be based on the alpha spending function concept, according to Lan and DeMets, and will employ O'Brien-Fleming Z-test boundaries, which are very conservative early in the trial. For the first interim analysis the efficacy stopping rule would require an extremely low P value (P< 0.000015). For the second interim analysis P< 0.003 will be taken as efficacy stopping rule. For the third interim analysis P< 0.02 will be taken as efficacy stopping rule. Investigators will be kept blind to the interim analysis results.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of SCD based on sickle cell tests and hemoglobin electrophoresis.
* Age 18 to 60 years
* Acute onset of painful crises, defined as having an onset within 7 days

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Altered mental status
* Body mass index greater than 40 kg/m2
* Patients with significant neurological disease
* Seizures
* Acute head injury
* Acute eye injury
* Patients with high intra-cranial tension
* Patients with known psychiatric disorders
* Patients with significant cardiac diseases
* Arrhythmias
* Patients with significant pulmonary diseases rather than acute chest syndrome
* Patients with significant renal disease (BUN/creatinine ratio < 25)
* Patients with significant hepatic disease (Child Pugh class B or C)
* Patients with significant endocrine disease
* Known allergy to phencyclidine derivatives
* Known allergy to ketamine
* Known allergy to morphine
* Sepsis
* Septic shock
* Patients required circulatory support
* Patients required ventilatory supports
* Alcohol abuse
* Drug abuse
* Patients with chronic pain status unrelated to SCD
* Patients receiving anti-convulsant medications
* Patients receiving anti-psychiatric medications.
* Patients with communication barriers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 278 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed SS Alshahrani, MD, Principal Investigator — King Fahad Hospital of the University -Imam Abdulrahman Bin Faisal University - (Dammam University)
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical plan, and results will be shared after publishing the manuscript. Currently, it is submitted and under peer review.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: for 5 years after completing the study
Access Criteria: Through direct contact with the Principal Investigator

REFERENCES:
- [Derived] Alshahrani MS, Asonto LP, El Tahan MM, Al Sulaibikh AH, Al Faraj SZ, Al Mulhim AA, Al Abbad MF, Al Nahhash SA, Aldarweesh MN, Mahmoud AM, Almaghraby N, Al Jumaan MA, Al Junaid TO, Al Hawaj FM, AlKenany S, ElSayed OF, Abdelwahab HM, Moussa MM, Alossaimi BK, Alotaibi SK, AlMutairi TM, AlSulaiman DA, Al Shahrani SD, Alfaraj D, Alhazzani W. Study protocol for a randomized, blinded, controlled trial of ketamine for acute painful crisis of sickle cell disease. Trials. 2019 May 27;20(1):286. doi: 10.1186/s13063-019-3394-4. PMID 31133061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completed
Period: Overall Study
Arm/Group | Morphine Group | Ketamine Group
Started (Completed) | 140 | 138 (Completed)
Completed (Completed) | 140 | 138 (Completed)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine Group | Ketamine Group | Total
Number analyzed (Participants) | 140 | 138 | 278
Age, Continuous [Median (Standard Deviation); unit: years] | 29.6 (7.9) | 29.1 (8.4) | 29.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 116
  Male | 82 | 80 | 162
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 140 | 138 | 278
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Saudi Arabia | 140 | 138 | 278
Numerical Pain Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Patients were asked to rate their pain at initial assessment within 30 minutes upon arrival, and the score was recorded by the bedside nurse.
  units on a scale | 8.7 (1.3) | 8.6 (1.3) | 8.6 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores
Description: Mean difference in the numerical pain rating scale score over 3 hours. Pain was measured on a scale from 0 (no pain) to 10 (the worst pain)
Time Frame: NPRS will be recorded every 30 minutes for a maximum of 180 minutes.
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Morphine Group | Ketamine Group
Number analyzed (Participants) | 140 | 138
score on a scale | 5.6 (1.90) | 5.7 (2.13)

2. Secondary Outcome: Length of Stay in ED
Description: Described as time elapsed from the start of study medication to the readiness for hospital discharge.
Time Frame: for 5 hours following admission to ED
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Morphine Group | Ketamine Group
Number analyzed (Participants) | 140 | 138
hours | 4.8 (2.47) | 4.7 (1.98)

3. Secondary Outcome: Cumulative Use of Opioid
Description: The cumulative use of opioid will be recorded during the ED stay
Time Frame: for 3 hours following admission to the ED
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Morphine Group | Ketamine Group
Number analyzed (Participants) | 140 | 138
mg/kg | 0.13 (0.11) | 0.07 (0.07)

4. Secondary Outcome: The Rate of Hospital Admission
Description: Number of admitted patients to the hospital after enrollment to study
Time Frame: within 3 hours following study enrollment
Population: intention to treat analysis (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Group | Ketamine Group
Number analyzed (Participants) | 140 | 138
Participants | 34 | 26

5. Secondary Outcome: Drug-related Adverse Effects
Description: flushing, hypotension, altered mental status, itching, paresthesia, respiratory depression, dizziness, nausea, vomiting
Time Frame: 3 hours following drug administration
Population: intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Morphine Group | Ketamine Group
Number analyzed (Participants) | 140 | 138
Participants | 3 | 8

ADVERSE EVENTS:
Time Frame: 180 minutes
Arm/Group | Morphine Group | Ketamine Group
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/138
Other Adverse Events (participants affected / at risk) | 3/140 | 8/138
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine Group (N=140) | Ketamine Group (N=138)
nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
dizziness (Ear and labyrinth disorders) | 3 (3) | 3 (3)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations included this being a single centre trial, thereby restricting the generalizability of the findings. Also, 180 minutes might be a short timeframe to assess impact of a study drug. Moreover, we calculated the use of a single low dose of ketamine that might be inadequate to provide our hypothesized superiority in the ketamine treated arm. Therefore, future studies

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT03431285/Prot_SAP_000.pdf
  • Informed Consent Form (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03431285/ICF_001.pdf